CLINICAL TRIAL: NCT06560450
Title: Research Report: CERITER Clinical Study - Stride One
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ceriter Nederland BV (Industry)
Collaborators: FRAME Jessa Ziekenhuis, Belgium (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVA-STRIDE-1-FRAME01
Record Dates: First submitted 2024-08-08; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: CVA (Cerebrovascular Accident)
Keywords: CVA (Cerebrovascular Accident); Gait rehabilitation; Gait analysis; Tele-rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Ten patients were offered therapy using Stride One for one week. Several measurements are performed before the start of the therapy, immediately after the end of the intervention period and 2 days after the end of the therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Real-time audio feedback (Other): Physiotherapist-defined real-time audio feedback
  Interventions: Device: Stride One

INTERVENTIONS:
Device: Stride One — Stride One is a smart insole that provides real-time audio feedback (cues) to the patient when performing a certain exercise. The goal of Stride One is to allow patients to practice walking more intensively and with higher quality during rehabilitation.

SUMMARY:
The goal of this clinical study is to investigate the short-term impact of the use of Ceriter Stride One on the quality of gait in patients rehabilitating after a cerebrovascular accident (CVA). Stride One is a smart insole that provides real-time audio feedback (cues) to the patient when performing a certain exercise.

The main questions it aims to answer are:

* Will patients with a CVA show a qualitatively better gait pattern after training with a Stride One insole?
* Can patients maintain this improvement in gait pattern without audio feedback at the end of the training?

Participants will

* Receive daily gait rehabilitation using Stride One for 1 week
* The quality of the gait pattern was evaluated at the beginning and at the end of the week, with and without the use of Stride One
* An additional evaluation was performed three to four days after the end of therapy without the use of Stride One
* Immediately after the end of the intervention week, the patient and the treating therapist were asked about their findings regarding the use of Stride One while walking

DETAILED DESCRIPTION:
Both therapist and patient reported an improvement in the quality of the foot roll-off pattern in 100% of cases. This improvement was also objectively determined in the data measured by Stride One, with an average of 8% improvement on Stride One general quality parameter, and an average of 25% improvement on Stride One specific quality parameter for the specific patient. Furthermore, 89% of patients indicate that using Stride One helps them to understand their physiotherapist better, and 67% of patients indicate that they can practice more and better with Stride One.

Practicing one week with Stride One generates a positive clinical impact on the gait pattern. A lasting improvement in the gait pattern without using Stride One, three to four days after the intervention, could not be demonstrated in this short time period. Further research is needed to evaluate the effect of Stride One after more long-term use.

Additional research questions are suggested.

ELIGIBILITY:
Inclusion Criteria:

* CVA, residentially admitted to the rehabilitation center in Herk-de-Stad, Belgium
* Older than 18 years of age
* Gait problems as a result of the CVA
* Able to walk safely and independently (possibly with a walking aid)
* Able to understand and sign an information and consent form

Exclusion Criteria:

* Severe cognitive problems (attention) that make it difficult to understand instructions or follow feedback
* Hearing problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Complete and correct foot roll-off | 1 week while daily therapy was given
  The first primary endpoint of the study is the complete and correct foot roll-off (detected and interpreted in the Ceriter platform). Stride One provides auditory feedback to the patient, stimulating the patient to achieve a good roll-off of the foot. For each step it measures whether a correct heel-strike, mid-stance and terminal stance are achieved. The aim of Stride One is to teach patients to place their feet correctly, in order to obtain a better roll- off, using positive audio feedback.
Changed walking speed/greater number of steps per minute | 1 week while daily therapy was given

SECONDARY OUTCOMES:
Improved functional tests: 5x sit-to-stand (seconds) | Before the start of the therapy, immediately after the end of the intervention period and 2 days after the end of the therapy
  • 3-minute walking test with audio feedback (distance in meter + roll-off pattern and Recording of auditory feedback via CERITER software), only at T1 and T2
Improved functional tests: 3-minute walking test without audio feedback | Before the start of the therapy, immediately after the end of the intervention period and 2 days after the end of the therapy
  Distance in meter + roll-off pattern via CERITER software
Improved functional tests: 3-minute walking test with audio feedback | Before the start of the therapy and immediately after the end of the intervention period
  Distance in meter + roll-off pattern and recording of auditory feedback via CERITER software
Subjective experiences: questionnaires | Post intervention, 2 days after end of the therapy
  Immediately after the end of the intervention week, the patient and the treating therapist were asked about their findings regarding the use of Stride One while walking.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Meyer, Study Director — Frame Jessa Ziekenhuis
Locations (1):
- Frame, Jessa Ziekenhuis, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khoo IH, Marayong P, Krishnan V, Balagtas M, Rojas O, Leyba K. Real-time biofeedback device for gait rehabilitation of post-stroke patients. Biomed Eng Lett. 2017 Jun 7;7(4):287-298. doi: 10.1007/s13534-017-0036-1. eCollection 2017 Nov. PMID 30603178
- [Background] Kwakkel G, Stinear C, Essers B, Munoz-Novoa M, Branscheidt M, Cabanas-Valdes R, Lakicevic S, Lampropoulou S, Luft AR, Marque P, Moore SA, Solomon JM, Swinnen E, Turolla A, Alt Murphy M, Verheyden G. Motor rehabilitation after stroke: European Stroke Organisation (ESO) consensus-based definition and guiding framework. Eur Stroke J. 2023 Dec;8(4):880-894. doi: 10.1177/23969873231191304. Epub 2023 Aug 7. PMID 37548025
- [Background] Kim J, Jung S, Song C. The Effects of Auditory Feedback Gait Training Using Smart Insole on Stroke Patients. Brain Sci. 2021 Oct 21;11(11):1377. doi: 10.3390/brainsci11111377. PMID 34827376

DOCUMENTS (1):
  • Study Protocol (2023-10-11): https://cdn.clinicaltrials.gov/large-docs/50/NCT06560450/Prot_000.pdf